CLINICAL TRIAL: NCT02618200
Title: Creation of a Multimodality Image Database (MRI + Ultrasound) for the Development of a Computer Aided Diagnostic (CAD) System in Patients With Prostate Cancer
Brief Title: Creation of an Image Database for the Development of a Computer Aided Diagnostic (CAD) System in Patients With Prostate Cancer
Acronym: Echo-CAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL15_0100
Record Dates: First submitted 2015-11-27; First posted 2015-12-01 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Computer-Aided Diagnosis
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3D prostate ultrasound (Experimental): 3D prostate ultrasound will be performed in patients the day before radical prostatectomy
  Interventions: Device: 3D prostate ultrasound

INTERVENTIONS:
Device: 3D prostate ultrasound

SUMMARY:
Prostate cancer is currently detected by ultrasound-guided biopsy. Computer-aided diagnostic (CAD) systems based on multiparametric MRI are now capable of detecting most aggressive cancer foci non-invasively, but additional progress is needed for the technique to be accepted in clinical practice. We hypothesize that combining MRI and ultrasound imaging can improve the detection of cancerous tumors. As a first step in this direction, we need to create a database with MR images, 3D ultrasound images, and corresponding histopathology results, in patients treated by radical prostatectomy for prostate cancer. This is the purpose of the present study.

In a later stage (outside the scope of this study), we will be learning how to combine these images to best recognize cancerous tumors, we will use that knowledge to develop a new CAD system, and we will assess the performance of the new CAD. We expect this future system to improve the detection of prostate cancer and to reduce the number of patients requiring biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred for radical prostatectomy
* Patient with multiparametric prostate MRI (3T) performed in our institution (Edouard Herriot Hospital) in the year preceding the surgery
* Informed consent signed
* Patient affiliated to the French Health Insurance system

Exclusion Criteria:

* History of prostatic surgery or radiation therapy (prostatic or pelvic)
* History of hormone therapy for prostate cancer
* Previous surgery of the abdomino-perineal region, or other contraindication for transrectal ultrasound
* Patient on protection of the court, under supervision or under trusteeship
* Inability to express a consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Obtention of 3D ultrasound images | the day before radical prostatectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot - Service Service de radiologie, Lyon, France

REFERENCES:
- [Result] Jaouen T, Souchon R, Moldovan PC, Bratan F, Duran A, Hoang-Dinh A, Di Franco F, Debeer S, Dubreuil-Chambardel M, Arfi N, Ruffion A, Colombel M, Crouzet S, Gonindard-Melodelima C, Rouviere O. Characterization of high-grade prostate cancer at multiparametric MRI using a radiomic-based computer-aided diagnosis system as standalone and second reader. Diagn Interv Imaging. 2023 Oct;104(10):465-476. doi: 10.1016/j.diii.2023.04.006. Epub 2023 May 20. PMID 37345961
- [Result] Couchoux T, Jaouen T, Melodelima-Gonindard C, Baseilhac P, Branchu A, Arfi N, Aziza R, Barry Delongchamps N, Bladou F, Bratan F, Brunelle S, Colin P, Correas JM, Cornud F, Descotes JL, Eschwege P, Fiard G, Guillaume B, Grange R, Grenier N, Lang H, Lefevre F, Malavaud B, Marcelin C, Moldovan PC, Mottet N, Mozer P, Potiron E, Portalez D, Puech P, Renard-Penna R, Roumiguie M, Roy C, Timsit MO, Tricard T, Villers A, Walz J, Debeer S, Mansuy A, Mege-Lechevallier F, Decaussin-Petrucci M, Badet L, Colombel M, Ruffion A, Crouzet S, Rabilloud M, Souchon R, Rouviere O. Performance of a Region of Interest-based Algorithm in Diagnosing International Society of Urological Pathology Grade Group >/=2 Prostate Cancer on the MRI-FIRST Database-CAD-FIRST Study. Eur Urol Oncol. 2024 Oct;7(5):1113-1122. doi: 10.1016/j.euo.2024.03.003. Epub 2024 Mar 16. PMID 38493072